CLINICAL TRIAL: NCT04674826
Title: A Randomized, Open-label, 2-period, 2-sequence Cross-over Trial to Compare the Pharmacokinetics of Tralokinumab of Two Presentations in Healthy Subjects
Brief Title: A Trial to Compare the Pharmacokinetics of Tralokinumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LP0162-1491
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TR (Test-Reference) (Experimental): Treatment period 1: 300 mg tralokinumab, single subcutaneous dose, 1 × X mL Device A (Test treatment, T) Treatment period 2: 300 mg tralokinumab, subcutaneous dose, 2 × Y mL Device B (Reference treatment, R)
  Interventions: Drug: Tralokinumab administered as 1 × X mL with Device A; Device: Tralokinumab administered as 2 × Y mL with Device B
- RT (Reference-Test) (Experimental): Treatment period 1: 300 mg tralokinumab, subcutaneous dose, 2 × Y mL Device B (Reference treatment, R) Treatment period 2: 300 mg tralokinumab, single subcutaneous dose, 1 × X mL Device A (Test treatment, T)
  Interventions: Drug: Tralokinumab administered as 1 × X mL with Device A; Device: Tralokinumab administered as 2 × Y mL with Device B

INTERVENTIONS:
Drug: Tralokinumab administered as 1 × X mL with Device A — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous (SC) administration
Device: Tralokinumab administered as 2 × Y mL with Device B — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous (SC) administration

SUMMARY:
The purpose of this trial is to compare the pharmacokinetics (PK), safety, tolerability and immunogenicity of a single dose of 300 mg tralokinumab administered as a 1 × X mL subcutaneous (SC) injection with Device A and 2 × Y mL consecutive SC injections with Device B.

DETAILED DESCRIPTION:
This is a single center, randomized, open label, 2 period, 2 sequence cross over trial designed to compare the PK and to evaluate the safety, tolerability and immunogenicity of 300 mg tralokinumab administered as a 1 × X mL SC injection with Device A (test treatment [T]) and 2 × Y mL consecutive SC injections with Device B (reference treatment [R]) in healthy subjects. Additionally, the experience of tralokinumab being administered with Device A compared to Device B will be evaluated.

After being informed about the study and the potential risks, all subjects giving written informed consent will be enrolled and randomized to 1 of 2 treatment sequences, Sequence TR or Sequence RT in a 1:1 ratio (i.e., subjects receive the 2 treatments in the specified order).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 to 55 years (both included) at the time of Screening.
* Female subjects of childbearing potential must use a highly effective form of birth control throughout the trial and at least for 16 weeks after last administration of the investigational medicinal product (IMP) and must have a negative serum pregnancy test at Screening.

Exclusion Criteria:

* Systemic (non biologic) or topical treatment within 21 days prior to first dose administration unless in the opinion of the Investigator the medication will not interfere with the trial procedures or compromise safety.
* Active tuberculosis or history of incompletely treated tuberculosis based on medical history or medical report.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at Screening, or the subject taking antiretroviral medications as determined by medical history and/or subject's verbal report.
* History of a clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to randomization.
* History of a helminth parasitic infection within 6 months prior to the date of informed consent that has not been treated with or has failed to respond to standard of care therapy.
* History of anaphylaxis or severe allergic reaction following any biologic therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration time curve from time 0 (pre dose) extrapolated to infinity (AUC0-inf) in each Treatment Period derived from all observed concentrations in the time period pre dose to 16 weeks post dose | In each Treatment Period pre-dose to 16 weeks post dose
Area under the serum concentration time curve from time 0 (pre dose) to time of last quantifiable concentration in each Treatment Period derived from all observed concentrations in the time period pre dose to 16 weeks post dose. | In each Treatment Period pre-dose to 16 weeks post dose
Observed maximum serum concentration (Cmax) in each Treatment Period derived from all observed concentrations in the time period pre dose to 16 weeks post dose | In each Treatment Period pre-dose to 16 weeks post dose

SECONDARY OUTCOMES:
Time corresponding to observed maximum serum concentration (tmax) | In each Treatment Period pre-dose to 16 weeks post dose
Terminal half life (t½) in each Treatment Period derived from all observed concentrations in the time period pre dose to 16 weeks post dose | In each Treatment Period pre-dose to 16 weeks post dose
Apparent total body clearance (CL/F), calculated as dose/AUC0-inf | In each Treatment Period pre-dose to 16 weeks post dose
  (AUC0-inf: Area under the serum concentration time curve from time 0 (pre dose) extrapolated to infinity)
Apparent volume of distribution based on terminal phase (Vz/F), calculated as t½/ln(2)*CL/F | In each Treatment Period pre-dose to 16 weeks post dose
  (t½: Terminal half life; CL/F: Apparent total body clearance)
Number of treatment emergent adverse events (TEAEs) from Day 1 to Day 126 and of TEAEs from Day 127 to Day 239 (number of adverse events [AEs] emerging with each treatment) | Day 1 to Day 239
Presence of binding and neutralizing anti-drug antibodies (ADAs) at Days 1 (pre dose), 15, and 57 of Treatment Periods 1 and 2 and Day 239 | Day 1 to Day 239

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Pharma Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No